CLINICAL TRIAL: NCT00530023
Title: Pilot Study To Identify Effective Methods Of Training Pump Naïve Subjects To Use The Paradigm® 722 System And To Describe Clinical Effectiveness Compared To Subjects Continuing With Multiple Dose Injections (MDI) of Insulin
Brief Title: Feasibility Study for Training Pump Naïve Subjects To Use The Paradigm® System And Evaluate Effectiveness
Acronym: STAR2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Scott Lee, MD/ Director, Medical Affairs, Medtronic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEP195/Z25
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Results first posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-05

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. 722 (Active Comparator): 722 arm: MiniMed Paradigm REAL-Time System
  Interventions: Device: MiniMed Paradigm REAL-Time System
- 2. Multiple Daily Injections (MDI) (No Intervention): MDI arm: Continue with currently prescribed Multiple Daily Injection therapy. No change in treatment or regime for study.

INTERVENTIONS:
Device: MiniMed Paradigm REAL-Time System — MiniMed Paradigm 722 insulin pump The transmitter The sensor Paradigm Link Glucose Meter The ComLink
  Other Names: Medtronic MiniMed Paradigm insulin infusion pump (MMT-722); Transmitter (MMT-7701); Subcutaneous glucose sensor (MMT-7002); Medtronic CareLink Diabetes Management System (MMT-7334); Paradigm Link Glucose Meter (HMS-322200A)
  Arms: 1. 722

SUMMARY:
Feasibility study to compare the effectiveness of the Paradigm Sensor Augmented System versus subjects continuing to administer insulin in multiple dose injections. Evaluate the educational materials and time required for training subjects naïve to continuous subcutaneous insulin infusion (CSII) to use the Paradigm 722 REAL Time System in preparation for a large multi-center clinical trial

DETAILED DESCRIPTION:
Many subjects with Type 1 diabetes continue to manage their disease utilizing multiple daily injections, but despite frequent blood glucose checks, are unable to control their glycemic variability or lower their A1C levels. The MiniMed Paradigm REAL-Time System transmits sensor glucose values to the insulin pump every 5 minutes, allowing users to view their current glucose values as well as glycemic excursions and trends over a 24-hour period. The System will also alert users of high and low glucose levels, allowing subjects and their clinicians to make carefully monitored modifications to therapy. Additionally, data can be uploaded from the monitor into a personal computer, allowing the subject and clinician to see a complete picture of trends over time.

Subjects learning this technology would require a new approach to training if they were to master operation of an insulin pump, make effective use of the sensor technology and understand the complete picture provided by the software component. Subjects will be trained to first use the insulin pump, add the sensor and then utilize the software and the effectiveness of the training methods and timing will be measured using questionnaires designed to evaluate understanding of the device, Self Efficacy and User Acceptance. The group wearing the System will also be compared to subjects that continue on their current MDI therapy over a 15-week time period.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 18 - 70 years of age (inclusive)
* Subject is diagnosed with Type 1 Diabetes Mellitus as determined by the Investigator.
* Diabetes is diagnosed > (greater or equal to) six (6) months prior to study entry.
* A1C > 7.5% (greater than or equal to) as measured by the Central Laboratory at Screening Visit 1.
* Subject currently requires insulin administration by injection > (greater or equal to) three (3) times daily.
* Subject is currently (over past 3 months) performing an average of four (4) blood glucose measurements per day, as determined and documented by the investigator
* Subject has been treated in the investigator's practice or in a referring endocrinologist's practice for at least 6 months prior to the study
* Subject is fluent in speaking, understanding, and reading English.
* Subject is able and willing to perform the study procedures and agrees to wear sensors at least five (5) days per week (722 Arm only) during the study period.
* Subject is able to use the study devices (722 Arm only) as labeled
* Subject has reviewed and signed the Informed consent, HIPPA Authorization, and California Experimental Subject's Bill of Rights (California only).
* Subject has the capability to upload their insulin pumps or glucose meters every two weeks; access to the Internet and specific computer system requirements are necessary to participate in the study

Exclusion Criteria:

* Subject is pregnant or planning to become pregnant during the course of the study.
* Subject has a history of tape allergies that have not been resolved.
* Subject self-reports any skin abnormality (i.e. psoriasis, rash, and staphylococcus infection).
* Subject has any additional condition(s) (medical, social, or psychosocial) that in the Investigator's opinion would warrant exclusion from the study or prevent the subject from completing or complying with the study requirements.
* Subject is currently or within past 4 weeks participated in an investigational study (drug or device).

Subject has a history of tape allergies that have not been resolved.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Lee, MD, Study Director — Medtronic Diabetes
Locations (2):
- United States (2):
  - Diabetes Treatment Center, Loma Linda University, Loma Linda, California
  - Portland Diabetes & Endocrinology, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Groups:
- 722 Sensor Augmented Insulin Pump: 722 MiniMed Paradigm REAL-Time System
- Multiple Daily Injections (MDI): Continue with current Multiple Daily Injection therapy
Period: Overall Study
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI)
Started | 14 | 15
Completed | 14 | 14
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI) | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 11 | 24
  >=65 years | 1 | 4 | 5
Age Continuous [Mean (Standard Deviation); unit: years] | 45.1 (12.59) | 49.7 (13.51) | 47.4 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 10 | 16
  Male | 8 | 5 | 13
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in A1C From Baseline to Week 15
Description: Change in A1C measured from Baseline to week 15 will be compared. A1C measured as percent of glycated hemoglobin using a standardized assay for all subjects.
Time Frame: Baseline and 15 weeks
Measure: Mean (Standard Deviation); unit: percent glycated hemoglobin
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 14 | 14
percent glycated hemoglobin | -1.7 (0.96) | -1.0 (0.97)

2. Secondary Outcome: Incidence of Severe Hypoglycemia Events Baseline to Week 15
Description: The total number of severe hypoglycemia events, defined as episodes requiring assistance from another person (i.e., subject is unable to treat self and requires carbohydrate or glucagon or other resuscitative actions) compared between the two study arms from Baseline to Week 15.
Time Frame: Baseline and 15 weeks
Measure: Number; unit: number of events
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 14 | 15
number of events | 0 | 1

3. Secondary Outcome: Blood Glucose Monitoring System - Ratings Questionnaire (BGMS-RQ) Assessed at Baseline and Week 15
Description: Questionnaire measuring overall satisfaction with the relevant blood glucose monitoring system. Assessed at Baseline and Week 15 and compared between arms. Likert scale used with responses graded as the lowest number being the least acceptable and the highest number the most acceptable. The scoring was then transformed to a 0 - 100 scale again with the higher number representing the most acceptable response.
Time Frame: Baseline and 15 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 14 | 14
Scores on a scale | 73.8 (26.7) | 41.0 (30.9)

4. Secondary Outcome: Insulin Delivery System - Ratings Questionnaire (IDS-RQ) Assessed at Baseline and Week 15
Description: Questionnaire measuring overall satisfaction with the relevant insulin delivery system. Assessed at Baseline and Week 15 and compared between arms. Likert scale used with responses graded as the lowest number being the least acceptable and the highest number the most acceptable. The scoring was then transformed to a 0 - 100 scale again with the higher number representing the most acceptable response.
Time Frame: Baseline and 15 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 14 | 14
Scores on a scale | 83.3 (21.7) | 33.3 (22.6)

5. Secondary Outcome: Hypoglycemia Fear Scale (HFS) Assessed at Baseline and Week 15
Description: Questionnaire evaluating change in the subjects' fear of potential hypoglycemia events assessed Week 15 and compared between arms. Likert scale of 0 - 4 used with responses graded as the lowest number being the most acceptable and highest number the least acceptable. The questionnaire has two sections, Behavior and Worry with a maximum possible score of 60 for Behavior (15 X 4) and 72 for Worry (18 X 4). The total combined scoring of these two sections was then assessed at Baseline and Week 15 and the change from Baseline to Week 15 for each arm reported as the end of study result.
Time Frame: Baseline and 15 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI)
Number analyzed (Participants) | 14 | 14
Scores on a scale | -10.57 (17.30) | -17.79 (19.99)

ADVERSE EVENTS:
Time Frame: 15 weeks
Description: Subject workbooks assessed at each visit. Discussion regarding SAE or AEs at each visit with reminders to call study personnel if SAE occured.
Arm/Group | 722 Sensor Augmented Insulin Pump | Multiple Daily Injections (MDI)
Serious Adverse Events (participants affected / at risk) | 1/14 | 3/15
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 722 Sensor Augmented Insulin Pump (N=14) | Multiple Daily Injections (MDI) (N=15)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Food Poisening (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less